CLINICAL TRIAL: NCT07115940
Title: Medical Management With Endovascular Thrombectomy Versus Medical Management Alone in Patients Presenting Beyond 24 Hours of Last Known Well - SELECT LATE Trial
Brief Title: Medical Management With Endovascular Thrombectomy Versus Medical Management Alone in Patients Presenting Beyond 24 Hours of Last Known Well
Acronym: SELECT LATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amrou Sarraj (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Amrou Sarraj, Professor of Neurology at the CWRU School of Medicine, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20250993; G250153 (Other: US Food and Drug Administration - CDRH)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
Keywords: Endovascular Thrombectomy; Mechanical Thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Practice Management, Medical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Medical Management with Endovascular Thrombectomy (Experimental): Medical management with endovascular thrombectomy (EVT) - EVT will be provided in addition to medical management and is a procedure to remove a thrombus in one of the brain arteries that is obstructing the blood flow. Removing this occlusion results in restoration of blood flow to ischemic brain tissue and salvage of the parts that are still viable, which is expected to improve functional outcomes. Endovascular thrombectomy procedure will be performed using stent retrievers, aspiration devices or combination approach at the discretion of the treating physician, using devices approved by the local regulatory authority. For patients treated in the United States of America, only US Food and Drug Administration-approved neurothrombectomy devices can be used.
  Interventions: Device: Endovascular Thrombectomy; Other: Medical Management
- Medical Management without Endovascular Thrombectomy (Active Comparator): Medical management without endovascular thrombectomy comprises various measures to prevent further deterioration, enhance patients' outcomes and prevent occurrence of a secondary stroke in short and long term. This includes 1) evidence-based practices for blood pressure management 2) Neurocritical care monitoring with appropriate osmotic therapy and neurosurgical interventions such as hemicraniectomy for management of cerebral edema that occurs due to infracted brain tissue based on local institutional protocol, 3) stroke etiology identification by requisite neurology , cardiology, immunology evaluations and 4) short and long-term strategies for secondary stroke prevention, including anticoagulation, antiplatelet therapy, medical optimization and modification of stroke risk factors such as hypertension, hyperlipidemia, diabetes and other potential comorbidities.
  Interventions: Other: Medical Management

INTERVENTIONS:
Device: Endovascular Thrombectomy — EVT will be provided in addition to medical management and is a procedure to remove a thrombus in one of the brain arteries that is obstructing the blood flow and is responsible for the occurrence of stroke. Removing this occlusion results in restoration of blood flow to ischemic brain tissue and salvages the parts that are still viable, which is expected to improve functional outcomes. Endovascular thrombectomy procedure will be performed using stent retrievers, aspiration devices or combination approach at the discretion of the treating physician, using devices approved by the local regulatory authority. For patients treated in the United States of America, only US Food and Drug Administration-approved neurothrombectomy devices can be used.
  Arms: Medical Management with Endovascular Thrombectomy
Other: Medical Management — Medical management comprises various measures to prevent further deterioration, enhance patients' outcomes and prevent occurrence of a secondary stroke in short and long term. This includes 1) evidence-based practices for blood pressure management 2) Neurocritical care monitoring with appropriate osmotic therapy and neurosurgical interventions such as hemicraniectomy for management of cerebral edema that occurs due to infracted brain tissue based on local institutional protocol, 3) stroke etiology identification by requisite neurology , cardiology, immunology evaluations and 4) short and long-term strategies for secondary stroke prevention, including anticoagulation, antiplatelet therapy, medical optimization and modification of stroke risk factors such as hypertension, hyperlipidemia, diabetes and other potential comorbidities.

SUMMARY:
SELECT LATE trial aims to evaluate if addition of endovascular thrombectomy to medical management in patients presenting with acute ischemic stroke and a proximal large vessel occlusion in the anterior circulation between 24 and 72 hours of stroke onset results in achieving better functional outcomes (measured using modified Rankin Scale Scores) at 90-day follow-up (± 15 days).

DETAILED DESCRIPTION:
SELECT LATE is a prospective, phase III, randomized, international, multicenter, assessor-blinded controlled trial evaluating if addition of endovascular thrombectomy to medical management in patients presenting with acute ischemic stroke and a proximal large vessel occlusion in the anterior circulation between 24 and 72 hours of stroke onset results in achieving better functional outcomes (measured using modified Rankin Scale Scores) at 90-day follow-up (± 15 days).

Patients with the final diagnosis of an acute ischemic stroke due to a large vessel occlusion in the internal carotid artery (ICA) or M1 segment of the middle cerebral artery (MCA), who present between 24-72 hours of when they were last known to be well and meet neuroimaging eligibility criteria [Non-contrast CT ASPECTS 3-10 and Ischemic core volume ≤150ml] will be randomized in a 1:1 ratio to thrombectomy plus medical management vs medical management alone. Patient assessments will be made at baseline, 24 hours post-randomization, discharge, 90 days and 1 year.

The primary endpoint is the Modified Rankin Scale (mRS) score at 90 (+/- 15) days. The primary outcome is a shift on 90-day mRS scores, with scores of 5 (severe disability requiring constant care) and 6 (death) merged to avoid considering a shift from 6 to 5 as an improvement. Secondary outcomes include functional independence (mRS score of 0-2), Utility weighted mRS, and Quality of Life measures. Safety outcomes include mortality, severe disability or death (mRS 5-6), incidence of symptomatic intracranial hemorrhage (sICH per SITS-MOST); and Imaging outcomes include infarct volume on MRI diffusion-weighted imaging (DWI) sequence (or CT if MRI is not feasible) 24-72 hours after randomization.

A maximum of 408 patients will be randomized across the study sites. Online randomization with Common Scale-Minimum Sufficient Balance algorithm will be used to balance the distribution of important variables. Interim analyses will be conducted at 136 and 272 patients, at which time the study may stop for efficacy or futility.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Adults (18-85* years) with the final diagnosis of an acute ischemic stroke$
* NIHSS ≥ 6
* Time from last-known-well to randomization >24 - 72 hours
* Pre-stroke modified Rankin Scale score of 0-1
* Eligible for thrombectomy and medical management
* Signed Informed Consent obtained
* Subject willing to comply with the protocol follow-up requirements
* Anticipated life expectancy of at least 3 months *Inclusive of both 18 and 85 years of age (i.e. up to 86th birthdate). $Subacute presentation - In-hospital stroke admissions with fluctuating clinical symptoms for patients who presented to EVT centers within 24 hours of when they were last known well will not be eligible for the trial.

General Exclusion Criteria

* Current participation in another investigational interventional drug or device study.
* Baseline Platelet count <100,000/μl

Imaging Inclusion Criteria

* Proven large vessel occlusion in ICA or MCA-M1 occlusion (carotid occlusions can be cervical or intracranial, with or without tandem MCA lesions), as determined by MR Angiography (MRA) or CT Angiography (CTA)
* CT ASPECTS 3-10
* CT Perfusion ischemic core (rCBF <30%)# volume ≤150 ml OR MR Diffusion ischemic core (ADC <620x10-6 mm2/s)# volume ≤150ml #If the perfusion software at enrollment center uses another threshold/measure to define ischemic core, please use that measure to assess ischemic core criteria.

Imaging Exclusion Criteria

* Evidence of intracranial tumor (except small meningioma <3cm without signs of edema or inflammation), acute intracranial hemorrhage, or arteriovenous malformation
* Significant mass effect, defined as midline shift (>3mm) using foramen of monroe (anterior margin of third ventricle) as the marker for midline instead of septum pellucidum AND/OR Effacement of sulci in contralateral hemisphere
* Evidence of internal carotid artery dissection that is flow limiting or aortic dissection
* Intracranial stent implanted in the same vascular territory that precludes the safe deployment/removal of the neurothrombectomy device
* Acute symptomatic arterial occlusions in more than one vascular territory confirmed on CTA/MRA (e.g., bilateral MCA occlusions, or an MCA and a basilar artery occlusion).
* Any signs of established infarct, demarcating hypodensity and area of cerebral edema on non-contrast CT
* CT ASPECTS 0-2
* CT Perfusion ischemic core (rCBF <30%)# volume >150 ml OR MR Diffusion ischemic core (ADC <620x10-6 mm2/s)# volume >150ml #If the perfusion software at enrollment center uses another threshold/measure to define ischemic core, please use that measure to assess ischemic core criteria.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
The distribution of the modified Rankin Scale score | 90 days ± 15 days
  The modified Rankin Scale (a 7-point scoring system, 0 indicates no residual stroke symptoms and 6 represents death) is assessed through patient/caregiver interview by trained and certified raters. The modified Rankin Scale score is the standard FDA-recognized measure of stroke outcome, used in clinical trials testing acute stroke therapies.

SECONDARY OUTCOMES:
Utility-weighted modified Rankin Scale scores | 90 days ± 15 days
  The Utility-Weighted Modified Rankin Scale (UW-mRS) is an advancement in the assessment of disability and functional independence for patients with neurological conditions. By incorporating patient preferences, it complements the traditional Modified Rankin Scale (mRS) by capturing individual preferences for specific health states. UW mRS is calculated by incorporating responses from the EuroQol-5 Dimension (EQ-5D) questionnaire, with a maximum score of 10 and minimum score of 0 and higher score indicating better functional status.
Domain-specific scores for NeuroQoL | 90 days ± 15 days
  The Neuro-Quality of Life (Neuro-QoL) measurement system evaluates health-related quality of life (HRQoL) in patients with neurological conditions through patient-reported outcomes, incorporating the impact of diseases and treatments on patients' daily lives and well-being. Neuro-QoL comprises item banks in Motor, Social, Cognitive and Depression modules. Responses to questions are converted into T-scores ranging from 0 to 100, with higher scores for Motor, Social and Cognitive domains indicating better quality of life and higher scores for depression domain indicating worse quality of life.
Functional independence (mRS 0-2) | 90 days ± 15 days
  Functional independence is identified by pooling all patients achieving a) no stroke deficits (mRS of 0), b) minimal stroke deficits without any functional limitations (mRS of 1) and c) functional limitations that do not interfere with independent living (mRS of 2) and illustrates being able to execute all day to day activities required for independent living, including bathing and dressing, cooking, grocery shopping and handling finances, with or without some degree of stroke deficits present.
The distribution of the modified Rankin Scale score | 1 year ± 30 days
  The modified Rankin Scale (a 7-point scoring system, 0 indicates no residual stroke symptoms and 6 represents death) is assessed through patient/caregiver interview by trained and certified raters. The modified Rankin Scale score is the standard FDA-recognized measure of stroke outcome, used in clinical trials testing acute stroke therapies.
Functional independence (mRS 0-2) | 1 year ± 30 days
  Functional independence is identified by pooling all patients achieving a) no stroke deficits (mRS of 0), b) minimal stroke deficits without any functional limitations (mRS of 1) and c) functional limitations that do not interfere with independent living (mRS of 2) and illustrates being able to execute all day to day activities required for independent living, including bathing and dressing, cooking, grocery shopping and handling finances, with or without some degree of stroke deficits present.
Utility-weighted modified Rankin Scale scores | 1 year ± 30 days
  The Utility-Weighted Modified Rankin Scale (UW-mRS) is an advancement in the assessment of disability and functional independence for patients with neurological conditions. By incorporating patient preferences, it complements the traditional Modified Rankin Scale (mRS) by capturing individual preferences for specific health states. UW mRS is calculated by incorporating responses from the EuroQol-5 Dimension (EQ-5D) questionnaire, with a maximum score of 10 and minimum score of 0 and higher score indicating better functional status.
Domain-specific scores for NeuroQoL | 1 year ± 30 days
  The Neuro-Quality of Life (Neuro-QoL) measurement system evaluates health-related quality of life (HRQoL) in patients with neurological conditions through patient-reported outcomes, incorporating the impact of diseases and treatments on patients' daily lives and well-being. Neuro-QoL comprises item banks in Motor, Social, Cognitive and Depression modules. Responses to questions are converted into T-scores ranging from 0 to 100, with higher scores for Motor, Social and Cognitive domains indicating better quality of life and higher scores for depression domain indicating worse quality of life.

OTHER OUTCOMES:
Symptomatic Intracerebral Hemorrhage (sICH) | 24 hours ± 6 hours
  Symptomatic Intracerebral Hemorrhage (sICH) is defined using SITS-MOST criteria (worsening of 4 or more points in NIH stroke scale score associated with parenchymal hematoma involving >30% of the infarct bed or remote parenchymal hematoma or symptomatic subarachnoid hemorrhage).
Presence and type of Intracerebral Hemorrhage (ICH) | 24 hours ± 6 hours
  defined using Heidelberg classification
Mortality | 90 days ± 5 days
  death by the time of follow-up completion
Number of patients receiving surgical decompression for cerebral edema | 7 days
  Number of patients receiving any surgical intervention to relieve cerebral edema and prevent/reduce its undesired effects

CONTACTS AND LOCATIONS:
Overall Officials: Amrou Sarraj, MD, Principal Investigator — University Hospitals

IPD SHARING:
Plan to Share IPD: Yes
De-identified Individual patient-level data will be submitted to repository designated by the funding agency.